CLINICAL TRIAL: NCT03185533
Title: Reducing Length of Stay in the Emergency Department: Analyzing the Factors and Quality Improvement Interventions
Brief Title: Reducing Length of Stay in the Emergency Department
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, Wan-Ching Lien, Director, Department of Emergency Medicine, NTUH Hsin-Chu branch, National Taiwan University Hospital Hsin-Chu Branch
Other Study IDs: 105-061-E
Record Dates: First submitted 2017-06-04; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Length of Stay
MeSH Terms: interventions — Quality Improvement; Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- to reduce ED length of stay: to reduce ED length of stay to lessen ED crowding by using Lean-sigma management and quality improvement interventions including reducing boarding time and medical decision time.
  Interventions: Behavioral: Quality improvement (QI) interventions

INTERVENTIONS:
Behavioral: Quality improvement (QI) interventions — 1. The ED admissions exhibited prolonged length of stay.
  2. The Interventions for Reducing Medical Decision Time:
  1. The ED director created QI education sessions and reported monthly QI outcomes.
  2. The ED nurses reported the current number of ED admission patients twice a day to the director. The director summarized the bed requests to the administrative personnel.
  3. The nurses reported the in-scene complicated cases to the ED director. The director would give an assistance in managing these cases.
  3. The Interventions for Reducing Boarding Time
  1. The ED patients could be admitted before 8 a.m. if the bed was vacant.
  2. The ED director initiated an on-line meeting at 8 a.m. and 4 p.m.
  3. Monthly QI outcomes were reported in the hospital affairs meeting.

SUMMARY:
Emergency department (ED) crowding has become an international challenge in the recent decades.

Length of stay (LOS) is a useful marker to monitor ED crowding. Searching for the possible causes and reducing barriers may have the greatest impact on EDLOS.

Therefore, the investigators assembled a multidisciplinary team for improvement of the ED process, to undergo assessments of ED patient flow with the spirit of lean-sigma methodologies. The objectives of this study were to evaluate a Lean-sigma-based initiative to lessen EDLOS.

DETAILED DESCRIPTION:
Lean aims to smooth out the workflow and to eliminate wastes. In the ED settings, lean principles can display the process of the ED patient flow. Six sigma, a complementary strategy, has the merit to compensate the potential weakness of Lean through a data-driven process. Currently, a combination of Lean and Six sigma methodologies develops to solve the problems of workflow.

It became clear that concurrent multifaceted interventions were needed to reduce EDLOS. Therefore, the investigators assembled a multidisciplinary quality improvement team for improvement of the ED process, to undergo assessments of ED patient flow with the spirit of lean-sigma methodologies. The objectives of this study were to evaluate a Lean-sigma-based initiative to lessen EDLOS.

ELIGIBILITY:
Inclusion Criteria:

* the patients were registered in the ED from Jan, 2015 to Dec, 2015.

Exclusion Criteria:

* the patients were excluded because of left without seeing a physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients were registered in the ED of the Hsin-Chu branch from Jan, 2015 to Dec, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 72000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
length of stay for ED admissions. | 12 months
  Length of stay was defined as the time from patient registration to leaving the ED.

SECONDARY OUTCOMES:
boarding time for ED admissions | 12months
  Boarding time was defined as the time from decision for admission to leaving the ED.
decision time for ED admissions | 12 months
  Decision time was defined as the time from patient registration to decision for disposition.
the percentage of LOS over 24 hours in all ED patients. | 12 months
  The percentage was defined as patients staying at the ED over 24 hours/total ED visits.

IPD SHARING:
Plan to Share IPD: Yes